CLINICAL TRIAL: NCT04234269
Title: Cultural Adaptation and Turkish Version of Physical Activity Scale for Individuals With Physical Disabilities in Individuals With Spinal Cord Injury: a Reliability and Validity Study
Brief Title: Physical Activity Scale in Individuals With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Other Study IDs: 006
Record Dates: First submitted 2020-01-02; First posted 2020-01-21 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment Group: Individuals with spinal cord injury. There is one group.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Evaluation forms will be applied to the patients who meet the inclusion criteria by face to face interview method.The sociodemographic information of the patients and the time taken to answer the questions in the questionnaires will vary according to each patient, but will take approximately 45 minutes. The second interview will be conducted with the patients for test-retest application at 1 week intervals.

SUMMARY:
The aim of this study was to improve the cultural adaptation and Turkish version of the The Physical Activity Scale for Individuals With Physical Disabilities (PASIPD) and to investigate the validity and reliability of the Turkish version of PASIPD in individuals with spinal cord injury. PASIPD, which consists of 13 questions, will be adapted to Turkish by translation and back translation method. The study included 47 wheelchair-dependent patients over the age of 18 who were able to read and write Turkish (26 females, 21 males). In order to determine the reliability and internal consistency of PASIPD, item-total correlation, if item deleted cronbach alpha coefficient and cronbach alpha coefficient of the whole scale will be calculated. Test-retest method will be used for the stability of the scale. In the test-retest method, the scale will be re-applied to the same people with 7-day intervals. Pearson correlation analysis will be performed between the first test and the second test total and sub-parameters after 1 week. Test-retest reliability will be determined using the intraclass correlation coefficient (ICC). In the validity test of PASIPD; construct validity and criterion validity will be used. Test of construct validity; factor analysis and convergent and discriminant validity methods. The Barthel Index of Activities of Daily Living and Functional Independence Measure (FIM); World Health Organization Quality of Life Scale Abbreviated Version (WHOQOL-BREF), Nottingham Health Profile (NHP) and Craig Handicap Assessment and Reporting Technique (CHART-SF) will be used to convergent and discriminant validity. Manual Wheelchair Propulsion Tests will be used to demonstrate criterion validity.

ELIGIBILITY:
Inclusion Criteria:

* Classified as group A, B, C or D according to American Spinal Injury Association (diagnosed with spinal cord injury),
* Fully or partially wheelchair dependent
* Over 18 years old
* Willing to research,
* Can read and write and read and write in Turkish
* Patients without cognitive impairment.
* Having the upper extremity muscle strength required for wheelchair use

Exclusion Criteria:

* Reluctant and unwilling to research,
* Having any progressive discomfort
* Bed dependent,
* Patients with severe cognitive impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study will be made on Turkey Spinal Cord Injury Association in ages ranging from ages 18-75 enrolled 47 volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | 12 weeks
  Functional Independence Measure evaluates the daily living activities. It comprises 18 items; 13 motor items (self-care and locomotion) and five cognitive items (communication and cognition), each of which is scored on a seven-point scale. The motor and cognitive scores have been separated, and each score now has a range of 0-100. The total score ranges from 13 to 126. A lower score indicates a worse functional level.
The Barthel Index of Activities of Daily Living | 12 weeks
  The Barthel Index evaluates the activities of daily living. The total Barthel Index score ranges from 0-100. 0 represents full dependency, 100 represents full independence. A score above 60 indicates independence in daily living activities.
20 meters push test | 12 weeks
  It is the one of the Manual Wheelchair Propulsion Tests. Manual Wheelchair Propulsion Tests to evaluate participants' ability to use manual wheelchairs. Patients ride their wheelchairs as fast as they can on a 20-meter course. At this time, the evaluator records how many seconds the 20-meter course is completed.
slalom test | 12 weeks
  It is the one of the Manual Wheelchair Propulsion Tests. Manual Wheelchair Propulsion Tests to evaluate participants' ability to use manual wheelchairs. An 18-meter course; 3 cones at 3 meter intervals, 2 cones at 2 meter intervals, 2 cones at 1 meter intervals. Patients progress by making slalom between cones and come back by making slalom from the last cone. At this time, an evaluator records the number of seconds the track has been completed.
6 Minute Push Test | 12 weeks
  It is the one of the Manual Wheelchair Propulsion Tests. Manual Wheelchair Propulsion Tests to evaluate participants' ability to use manual wheelchairs. An eight-course track of 25 meters in length; in the middle and on both sides of the cones. Patients start in the middle of the course. It then moves quickly to the cone on the right or left edge and returns to the center of the track. At the next stage, it moves to the cone on the other side of the course and proceeds for 6 minutes. At this time, an evaluator will record the number of meters traveled in 6 minutes.
Nottingham Health Profile | 12 weeks
  It measures the quality of life. The questionnaire consists of 38 items and evaluates six dimensions related to health status. Questions are answered as yes or no. Each section is scored between 0-100. 0 indicates the best health status, 100 indicates the worst health status.
World Health Organization Quality of Life Scale Abbreviated Version | 12 weeks
  World Health Organization Quality of Life Scale Abbreviated Version evaluates the quality of life. It consists of 4 sections: physical health (seven items), psychological health (six items), social relations (three items), environment (eight items), and two additional items that score the perception of health and quality of life.The minimum score is 0 and the maximum score is 100. Higher score shows better result.
Craig Handicap Assessment and Reporting Technique. | 12 weeks
  Craig Handicap Assessment and Reporting Technique evaluates the quality of life. The scale consists of 5 parts: physical independence, mobility, roles and activities, social integration, economic self-sufficiency. Each parameter is scored between 0-100. The higher the participation, the higher the score, the lower the disability. The maximum score of 100 represents the level of participation of the non-disabled person.
Physical Activity Scale for Individuals with Physical Disabilities | 12 weeks
  The Physical Activity Scale for Individuals with Physical Disabilities evaluates the physical activity level. It is a 13-item personal report form for the purpose of classifying daily living activities (items 1-6), domestic activities (items 7-12) and professional tasks (items 13) in the last seven days.The minimum score is 0 MET hr/d and the maximum score is 199.5 MET hr/d. Higher score shows better result.

CONTACTS AND LOCATIONS:
Locations (1):
- İstinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koce K, Atici E, Buran Cirak Y, Durustkan Elbasi N, Tutuneken YE. Cultural adaptation and Turkish version of Physical Activity Scale for Individuals with Physical Disabilities in individuals with spinal cord injury: a reliability and validity study. Disabil Rehabil. 2022 Oct;44(21):6414-6423. doi: 10.1080/09638288.2021.1964624. Epub 2021 Aug 20. PMID 34415222